CLINICAL TRIAL: NCT06410066
Title: Outcomes of Non-COVID-19 Critically Ill Patients With Hematologic Malignancies
Brief Title: Outcomes of Critically Ill Patients With Hematologic Malignancies
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ori Galante, senior physician, head of ECMO service SUMC, Soroka University Medical Center
Other Study IDs: 0038-20-SOR
Record Dates: First submitted 2024-05-02; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hematologic Malignancy
Keywords: intensive care unit; haematologic malignancy; mortality
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PATIENTS WITH HEMATOLOGIC MALIGNANCY aADMITTED TO THE ICU: all consecutive patients diagnosed with HM and admitted to both ICUs between January 2009 and December 2019.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The investigators sought to report the outcomes of patients with haematological malignancies admitted to the intensive care units and to define pre-intensive care units prognostic factors for in-hospital all-cause mortality.

In this retrospective, single-center study, all patients with haematologic malignancies admitted to intensive care units between 2009 and 2019 were included. The primary outcome was in-hospital mortality.

DETAILED DESCRIPTION:
The study was performed at the SUMC, an academic tertiary medical center serving the entire southern district of Israel. Our hospital operates two ICUs: an 8-bed medical ICU and a 16-bed surgical ICU. A senior intensivist and haematologist are available 24 hours every day for clinical decision-making at both units.

The investigators conducted a retrospective cohort study of all consecutive patients diagnosed with HM and admitted to both ICUs between January 2009 and December 2019. The inclusion criteria were a diagnosis of HM on admission or discharge from the ICU. Patients under 18 years of age or who were completely cured of malignancy for more than five years were excluded. Patients admitted to the ICU during the COVID-19 pandemic were also excluded to avoid biases caused by resource accessibility in terms of ICU beds and qualified teams.

The investigators collected data from the hospital's electronic medical records, including demographic data, medical history, and comorbidities, as coded by the International Classification of Diseases (ICD)-9.

Haematological malignancy diagnoses were categorized into five major groups: acute leukemia, aggressive non-Hodgkin lymphoma, Hodgkin lymphoma, multiple myeloma, and others. The remission status, post haematopoietic cell transplantation status (allogeneic or autologous), and date of the last chemotherapy or biological treatment were collected.

Clinical pre-ICU admission parameters, including vital signs, complete blood count, absolute neutrophil counts, lactate dehydrogenase (LDH) levels, liver enzymes, urea and creatinine levels, electrolytes, pH and lactate levels, and coagulation parameters, were recorded at ICU admission. Moreover, the ICU admission Sepsis-Related Organ Failure Assessment (SOFA) score 20 and the acute physiology and chronic health evaluation (APACHE) II severity of disease classification system 21 were recorded, to provide prognostic evidence-based references.

Clinical parameters during ICU admission included treatment with vasopressor medications, the level of respiratory support needed (nasal cannula/reservoir mask/noninvasive ventilation/invasive mechanical ventilation support), the need for renal replacement therapy, and liver dysfunction, defined by the elevation of liver enzymes and bilirubin.

The definition of organ dysfunction during ICU admission included the need for mechanical ventilation, vasopressor treatment, renal replacement therapy, elevated bilirubin >2 mg/dl or newly reduced left ventricular function (defined as an ejection fraction <30%).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HM on admission or discharge from the ICU

Exclusion Criteria:

* patients under 18 years of age patients who were completely cured of malignancy for more than five years patients admitted to the ICU during the COVID-19 pandemic

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients diagnosed with HM and admitted to both ICUs between January 2009 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
mortality | 30 day
  in hospital mortality

IPD SHARING:
Plan to Share IPD: No